CLINICAL TRIAL: NCT06641167
Title: Interest of Soft Point Anesthesia in Association With Locoregional Anesthesia in Arthroscopic Shoulder Surgery
Acronym: CAESAR
Status: Not yet recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-06-007
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Shoulder surgery — shoulder surgery by arthroscopic approach under locoregional anesthesia combining an interscalene block and a superficial cervical plexus block

SUMMARY:
This is a prospective, single-center, observational study. The inclusion period is set at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient informed about the study and who has not opposed the use of their personal medical data
* Patient scheduled for arthroscopic shoulder surgery

Exclusion Criteria:

* Allergy to local anesthetics or epinephrine
* Contraindications to Interscalene Block (e.g., respiratory disease, pneumothorax, pneumonectomy, phrenic or recurrent laryngeal nerve paralysis)
* Coagulation disorder
* Patients unable to understand the study information and objectives: dementia, psychosis, consciousness disorders, non-French-speaking patients
* Patients under legal protection measures (guardianship, curatorship) or deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population of patients undergoing shoulder surgery by arthroscopic approach under locoregional anesthesia combining an interscalene block and a superficial cervical plexus block (supraclavicular nerve)
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Soft point position | Hour 24
  The primary outcome is the position of the soft point in relation to the anesthetized area mapped by loco-regional anesthesia

SECONDARY OUTCOMES:
Incision pain | Hour 24
  Assessment of incision pain using a simple numerical scale (NRS) from 0 (no pain/not uncomfortable) to 10 (worst possible pain/most uncomfortable)
Postoperative pain | Hour 2
  Assessment of postoperative pain using a simple numerical scale (NRS) from 0 (no pain) to 10 (worst possible pain)
Postoperative pain | Hour 6
  Assessment of postoperative pain using a simple numerical scale (NRS) from 0 (no pain) to 10 (worst possible pain)
Postoperative pain | Hour 24
  Assessment of postoperative pain using a simple numerical scale (NRS) from 0 (no pain) to 10 (worst possible pain)
Sedative medication | Hour 24
  Amount of sedative medication administered
Analgesic consumption | Hour 24
  Amount of analgesics consumed within the 24 hours following surgery
Intervention duration | Hour 24
  Duration of the procedure and stay in the Post anesthesia care unit (the procedure duration is defined as the time between the start of the incision and the end of suturing)
Stay in the PACU duration | Hour 24
  Duration of the procedure and stay in the Post anesthesia care unit (the procedure duration is defined as the time between the start of the incision and the end of suturing)
Adverse events | Hour 24
  Perioperative and immediate postoperative adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé Claude Galien, Quincy-sous-Sénart, France

IPD SHARING:
Plan to Share IPD: No